CLINICAL TRIAL: NCT04753008
Title: Respiratory Effects of Dopamine in the Perioperative Care
Acronym: DOPHUMAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DOPHUMAN
Record Dates: First submitted 2021-02-05; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Dopamine; Bronchodilation; Heart; Surgery; Functional Disturbance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dopamine group (Experimental): Cardiac surgery patients receiving dopamine to support their cardiac function (as part of the routine post-operative care).
  Interventions: Drug: Dopamine administration
- Control group (No Intervention): Cardiac surgery patients receiving no positive inotrope drug.

INTERVENTIONS:
Drug: Dopamine administration — Administration of dopamine (3 mcg/kg/min) as part of cardiac support therapy after the cardiopulmonary bypass. Administration of dopamine is a subject of clinical decision based on the cardiovascular status of the patients.
  Arms: Dopamine group

SUMMARY:
Dopamine is frequently used as an inotropic drug to elevate cardiac output. In addition to the beneficial cardiac effect of this drug, the few previous studies addressing its ability to alter the airway tone reported controversial results.

Thus, the investigators aimed at clarifying the potential of dopamine to alter gas exchange outcomes and the airway tone in patients undergoing cardiac surgeries with cardiopulmonary bypass.

Blood gas parameters, airway resistance, tissue damping and tissue elastance will be measured in the patients before the CPB, immediately after CPB, and 5 min after administration of dopamine (3 mcg/kg/min).

The importance of the research is to reveal whether the beneficial mechanical changes after dopamine administrations are associated with improvements in gas exchange outcomes. Clarification of this research question have scientific relevance and may also improves patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Cardial surgery patients undergoing cardiopulmonary bypass procedures

Exclusion Criteria:

* Chronic respiratory diseases, elderly (>80 years)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-12-13 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Arterial oxygen partial pressure (PaO2) | 5 min after administration of dopamine
  Partial pressure of oxygen in the blood sample assessed by a blood gas analyser.
Arterial carbon dioxide partial pressure (PaCO2) | 5 min after administration of dopamine
  Partial pressure of carbon dioxide in the blood sample assessed by a blood gas analyser.
Lung mechanics | 5 min after administration of dopamine
  Airway resistance, lung tissue damping and lung tissue elastance obtained by forced oscillation technique.

SECONDARY OUTCOMES:
Capnography | 5 min after administration of dopamine
  Time capnography to obtain phase 3 and phase 2 slopes.
Intrapulmonary shunt | 5 min after administration of dopamine
  Intrapulmonary shunt obtained by the Berggren shunt equation from arterial and central venous blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Barna Babik, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No